CLINICAL TRIAL: NCT03630432
Title: A Pragmatic, Randomised, Controlled, Trial of the Effect of a Tailored Pulmonary Rehabilitation Package in Uncontrolled Asthma Associated With Elevated Body Mass Index
Brief Title: Pulmonary Rehabilitation for Uncontrolled Asthma Associated With Elevated BMI
Acronym: PRODA01
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GN16RM503
Record Dates: First submitted 2017-05-26; First posted 2018-08-14 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Asthma
Keywords: Severe; Difficult; Overweight and obese
MeSH Terms: conditions — Asthma; Lymphoma, Follicular; Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: Randomised, parallel, controlled study of 8 weeks pulmonary rehabilitation versus usual care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Immediate 8 week course of pulmonary rehabilitation
  Interventions: Behavioral: Pulmonary rehabilitation
- Group B (Placebo Comparator): Initial 8 weeks of usual care
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Pulmonary rehabilitation — The pulmonary rehabilitation course will be provided on a rolling basis and for each individual will be of 8 weeks duration including once weekly, 1.5 hour hospital sessions and encouragement to perform twice weekly home exercise sessions. Hospital sessions will include 1 hour of supervised exercise and 30 minutes education.
  Exercise Component: This will include a combination of aerobic, resistance and flexibility training.
  Educational Component will cover many topics including what is asthma, treatments and inhaler technique, self-management, importance of exercise and health promotion.
  On completion of the formal pulmonary rehabilitation course, participants will be encouraged to continue regular exercise sessions by accessing community based "Vitality Classes".
  Arms: Group A
Other: Usual Care — Usual Care
  Arms: Group B

SUMMARY:
Aim to evaluate the impact of a pulmonary rehabilitation (rehab) programme tailored and delivered to overweight and obese patients with difficult asthma on:

1. Asthma related quality of life (primary outcome) and asthma control (secondary outcome)
2. Treatment burden and healthcare usage (secondary outcomes)
3. Physical activity level, exercise tolerance, lung function and inflammation (secondary outcome)
4. Anxiety and depression (secondary outcome)

DETAILED DESCRIPTION:
Eligible individuals will be identified through Difficult Asthma Clinics or ward admissions. Those wishing to participate will receive an information sheet and be invited to provide written informed consent prior to commencing the study.

Baseline Visit

Measurements taken at the baseline visit will include:

Demographics - age, gender, smoking history (current, ex, none, years since stopped, pack years), age at asthma diagnosis, duration of asthma, atopy, co-morbidities (allergic/perennial rhinitis, nasal polyps, nasal surgery, eczema, gastro-oesophageal reflux disease (GORD), diabetes, hypertension, cardiac disease, osteopenia/osteoporosis etc), medications (inhaled/nebulised short acting beta2-agonists (SABA), inhaled and oral corticosteroids (OCS) etc), healthcare usage (oral corticosteroid boosts, unscheduled general practice (GP) or accident and emergency (A+E) attendances, hospital and intensive care unit (ICU) admissions in preceding year), weight, height and body mass index (BMI).

Questionnaires - Medical Research Council (MRC) dyspnoea scale, Asthma Control Questionnaire (ACQ6), Asthma Quality of Life Questionnaire (AQLQ), and Hospital Anxiety and Depression Scale (HAD).

Inflammatory - Blood eosinophils, Fraction of exhaled nitric oxide (FENO).

Lung Function - peak expiratory flow (PEF) (best of 3), Spirometry (pre- and post-bronchodilator).

Exercise tolerance - 6 minute walk test (6MWT) (practice test and repeat test), Modified Borg Dyspnoea Scale, pulse oximetry.

Physical Activity - actigraphy

Participants will be provided with a Personalized Asthma Management Plan, and Symptoms Diary that includes SABA use and other healthcare usage (OCS) boosts, unscheduled GP or A+E attendances, hospital and ICU admissions); inhaler technique will be corrected if necessary.

Participants will be randomized 1:1 to Group A and Group B. Group A will enter the 8 week pulmonary rehabilitation arm of the study immediately while Group B will enter the 8 week usual care arm. Group A will return for Visit 2 and Group B for Visit 1(2) at 8 weeks.

Measurements taken at Visits 1(2), 2. and 3 will include:

Demographics - medications (inhaled/nebulised short acting beta2-agonists (SABA), inhaled and oral corticosteroids etc), healthcare usage (OCS) boosts, unscheduled GP or A+E attendances, hospital and ICU admissions since last visit), weight, height, and BMI.

Questionnaires - MRC dyspnoea scale, Asthma Control Questionnaire (ACQ6), Asthma Quality of Life Questionnaire (AQLQ), and Hospital Anxiety and Depression Scale (HAD).

Inflammatory - Blood eosinophils, Fraction of exhaled nitric oxide (FENO).

Lung Function - PEF (best of 3), Spirometry (pre- and post-bronchodilator).

Exercise tolerance - 6 minute walk test, Modified Borg Dyspnoea Scale, pulse oximetry.

Physical Activity - actigraphy

After Visit 2, Group A will discontinue pulmonary rehabilitation; Group A will return for Visit 3 (48 weeks). Group B will enter the 8 week pulmonary rehabilitation arm and return for Visit 2 at 16 weeks; Group B will return for Visit 3 (56 weeks). Visits will be postponed by 4 weeks in the event of exacerbation or respiratory infection. Throughout the study period changes to asthma medications will be allowed as clinically indicated.

Pulmonary rehabilitation arm

The pulmonary rehabilitation course will be provided on a rolling basis and for each individual will be of 8 weeks duration including once weekly, 1.5 hour hospital sessions and encouragement to perform twice weekly home exercise sessions. Hospital sessions will include 1 hour of supervised exercise and 30 minutes education. Hospital sessions will run in Glasgow Royal Infirmary every Thursday morning with education (11:15-11:45) and exercise (12:00-13:00). Sessions will run with minimum 6 participants and aiming for 12-16.

Exercise Component: This will include a combination of aerobic, resistance and flexibility training. Participants will be screened prior to commencing exercise to confirm stability of asthma. Pre-exercise administration of bronchodilators (participant's own salbutamol inhaler) will occur and there will a gradual warm-up with stretches for 7 to 8 minutes. The prescribed training intensity will be defined by the exercise capacity during baseline 6MWT with progressive increase in repetitions. Nebulised salbutamol will be available in the venue. Individuals will then rotate through the following exercises:

12 leg extensions alternating right/left (R/L) +/- weights 12 arm weights (R/L together) 12 step ups Bike 12 Sit to stands 12 pole raises 12 knee lifts (alternating R/L) Walk

Educational Component: This will include the following topics:

What is asthma - and relation to physical activity Medications in asthma Recognizing warning signs, self management and personalized asthma action plans Inhaler technique and PEF recording Co-morbidities and asthma Dysfunctional breathing and breathing control exercises Anxiety management Relaxation Chest clearance Health promotion - smoking cessation, healthy eating etc Benefits of exercise and maintenance

On completion of the formal pulmonary rehabilitation course, participants will be encouraged to continue regular exercise sessions by accessing community based "Vitality Classes".

Usual care arm

During this 8 week period, individuals will be asked not to alter their physical activity level from baseline, and to continue their pre-study asthma management.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18-80 year (smokers, ex-smokers and non-smokers)
2. Confirmed asthma as per Global Initiative for Asthma (GINA) guidelines 2015[4] with characteristic symptoms and at least one of the following:

   * Airflow limitation - FEV1/FVC < 70% (at any time in the past) and 12% and 200ml increase in FEV1 in the preceding 5 years either:

     i. After inhaled/nebulised bronchodilator or 4+ weeks of anti- inflammatory treatment ii. Between visits
   * Positive bronchial challenge in the preceding 5 years:

   I. Histamine or methacholine provocation concentration causing a 20% drop in FEV1 (PC20) <8mg/ml ii. Provoking dose of mannitol required to cause a drop in FEV1 of 15% (PD15) mannitol <635mg
3. Difficult asthma defined as per Scottish Intercollegiate Guidelines Network(SIGN)/British Thoracic Society(BTS) guideline 2014 as persistent symptoms and/or frequent asthma attacks despite treatment at step 4 or step 5 with either:

   * ACQ6>1.5
   * ≥2 systemic corticosteroid boosts in previous year
   * ≥1 hospitalization in previous year
4. BMI≥25 kg/m2
5. MRC dyspnoea scale ≥3/5

Exclusion Criteria:

1. ICU admission +/- mechanical ventilation in the previous year for asthma exacerbation
2. Respiratory tract infection requiring antibiotics or asthma exacerbation requiring corticosteroid boost in preceding 4 weeks
3. Significant respiratory or other co-morbidity likely to influence the conduct of the study
4. Pregnancy and breast feeding
5. Severe and/or unstable cardiac disease
6. Impaired mobility that impacts on ability to participate in physical training
7. Recent (within the preceding 6 months) commencement of antifungal, biologic (omalizumab, lebrikizumab, mepolizumab) or Airsonett device; eligible if on treatment for >6months or discontinued >6 months ago.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2017-05-11 (Actual); Primary Completion 2019-05-10 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
AQLQ- Asthma quality of life questionnaire | 8 weeks
  change from week 0 to week 8 for pulmonary rehab vs usual care control group. AQLQ consists of 32 questions related to quality of life scored out of 7, and then averaged. Total score is out of 7 with 1 being the worst and 7 the best. There is also a score between 1 and 7 for 4 subscales which cover areas of symptoms, activity limitation, emotional function and environmental stimuli. These subscales are also averaged over a number of questions with 1 being worst and 7 best.

SECONDARY OUTCOMES:
AQLQ- asthma quality of life questionnaire | 8 weeks
  percentage with more than or equal to 0.5 point improvement from beginning to end of pulmonary rehab programme versus percentage in usual care control group. AQLQ consists of 32 questions related to quality of life scored out of 7, and then averaged. Total score is out of 7 with 1 being the worst and 7 the best. There is also a score between 1 and 7 for 4 subscales which cover areas of symptoms, activity limitation, emotional function and environmental stimuli. These subscales are also averaged over a number of questions with 1 being worst and 7 best.
ACQ6- asthma control questionnaire 6 | 8 weeks
  Change from week 0 to week 8 for pulmonary rehab vs usual care control group. ACQ6 comprises 6 questions scored out of 6 then averaged, value will range from 0-6, with 0 reflecting excellent asthma control and 6 very poor control.
ACQ6- asthma control questionnaire 6 | 8 weeks
  percentage with more than or equal to 0.5 point improvement from beginning to end of pulmonary rehab programme versus percentage in usual care control group. ACQ6 comprises 6 questions scored out of 6 then averaged, value will range from 0-6, with 0 reflecting excellent asthma control and 6 very poor control.
ACQ6- asthma control questionnaire 6 | 48 (or 56) weeks depending on group
  Change from baseline to end of study period. ACQ6 comprises 6 questions scored out of 6 then averaged, value will range from 0-6, with 0 reflecting excellent asthma control and 6 very poor control.
AQLQ | 48 (or 56) weeks depending on group
  Change from baseline to end of study period. AQLQ consists of 32 questions related to quality of life scored out of 7, and then averaged. Total score is out of 7 with 1 being the worst and 7 the best. There is also a score between 1 and 7 for 4 subscales which cover areas of symptoms, activity limitation, emotional function and environmental stimuli. These subscales are also averaged over a number of questions with 1 being worst and 7 best.
Change in treatment burden | 48 or 56 weeks
  Has there been a change in short acting beta agonist use, inhaled corticosteroid dose, maintenance prednisolone dose, frequency of prednisolone boosts; i.e. is the patient requiring any more or less treatment for asthma control than at baseline. This will be assessed by asking the patient and completing an asthma medication use treatment chart
Change in healthcare usage | 48/56 weeks
  Number of episodes of in scheduled care, including GP or A&E attendances, hospital and ICU admission. This will be compared to pre-trial episodes of the same.
Medical Research Council (MRC) dyspnoea score | 48/56 weeks
  Change in score on MRC dyspnoea scale. This is a score from 1-5 used to grade degree of breathlessness, 1 is the best result, 5 is the worst (most breathless)
Body mass index | 48/56 weeks
  Change in body mass index over study period, calculated using height in metres and weight in kilograms to give BMI in kg/m2
Inflammation | 48/56 weeks
  Changes in Blood eosinophils and FENO
Lung function | 48/56 weeks
  Change in forced expiratory volume in 1 second (FEV1) and forced vital capacity (FVC); lowest O2 saturation
Exercise tolerance | 48/56 weeks
  Change in 6MWT distance, modified Borg dyspnoea scale and lowest O2 saturation;
Physical activity | 48/56 weeks
  Change in actigraphy data
Hospital anxiety and depression scale | 48/56 weeks
  Change in score on HAD. This is a scale comprised of 14 questions where responses are graded from 0-3, with the responses then being totalled. A lower score is better, i.e. a higher score is indicative of more significant symptoms of anxiety and depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Glasgow Royal Infirmary, Glasgow, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ricketts HC, Sharma V, Steffensen F, Goodfellow A, Mackay E, MacDonald G, Buchan DS, Chaudhuri R, Cowan DC. A pragmatic randomised controlled trial of tailored pulmonary rehabilitation in participants with difficult-to-control asthma and elevated body mass index. BMC Pulm Med. 2022 Sep 24;22(1):363. doi: 10.1186/s12890-022-02152-2. PMID 36153525